CLINICAL TRIAL: NCT01779687
Title: Pharmacokinetic Drug Interaction Study Between Raltegravir and Atorvastatin (AVIATOR).
Brief Title: Pharmacokinetic Drug Interaction Study Between Raltegravir and Atorvastatin.
Acronym: AVIATOR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UMCNAKF-12.03
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2015-06

CONDITIONS: HIV; Hypercholesterolaemia
Keywords: pharmacokinetic; interaction; cholesterol; raltegravir; atorvastatin
MeSH Terms: conditions — Hypercholesterolemia | interventions — Raltegravir Potassium; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- raltegravir alone (Active Comparator): Raltegravir 400 mg BID for 7 days
  Interventions: Drug: raltegravir
- Atorvastatin alone (Active Comparator): Atorvastatin 20 mg QD for 7 days
  Interventions: Drug: Atorvastatin
- Raltegravir + atorvastatin (Experimental): Raltegravir 400 mg BID + Atorvastatin 20 mg QD for 7 days
  Interventions: Drug: raltegravir; Drug: Atorvastatin

INTERVENTIONS:
Drug: raltegravir — Raltegravir 400 mg BID for 7 days
  Other Names: raltegravir dosing for 7 days
  Arms: Raltegravir + atorvastatin; raltegravir alone
Drug: Atorvastatin — Atorvastatin 20 mg QD for 7 days
  Arms: Atorvastatin alone; Raltegravir + atorvastatin

SUMMARY:
Dyslipidemia is highly prevalent among patients with HIV infection and contributes to the increased cardiovascular disease risk in this patient population. Atorvastatin lowers plasma low-density lipoprotein (LDL) cholesterol levels and is used for prevention of artherosclerotic disease. Raltegravir, an HIV integrase inhibitor, could be one of the preferred antiretroviral agents in HIV patients with dyslipidemia because it has a beneficial lipid profile.

Theoretically, no clinically relevant drug interaction is expected between atorvastatin and raltegravir. However, atorvastatin and raltegravir share similar metabolic pathways which could be relevant in the occurrence of pharmacokinetic interactions. In order to be able to recommend raltegravir and atorvastatin concomitant use, a pharmacokinetic study in healthy volunteers is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 55 years at screening.
* Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to the first dosing
* Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry, haematology and urinalysis testing within 4 weeks prior to the first dose. Results of biochemistry, haematology and urinalysis testing should be within the laboratory's reference ranges. If laboratory results are not within the reference ranges, the subject is included on condition that the Investigator judges that the deviations are not clinically relevant. This should be clearly recorded.
* Subject has a normal blood pressure and pulse rate, according to the Investigator's judgement.

Exclusion Criteria:

* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Positive HIV test.
* Positive hepatitis B or C test.
* Pregnant female (as confirmed by an hCG test performed less than 4 weeks before day 1) or breast-feeding female. Female subjects of childbearing potential without adequate contraception, e.g. hysterectomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout the entire conduct of the study.
* Therapy with any drug (for two weeks preceding dosing), except for acetaminophen.
* Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disorders, renal and hepatic disorders, hormonal disorders (especially diabetes mellitus), coagulation disorders, musculoskeletal and connective tissue disorders.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* History of or current abuse of drugs, alcohol or solvents.
* Inability to understand the nature and extent of the study and the procedures required.
* Participation in a drug study within 60 days prior to the first dose.
* Donation of blood within 60 days prior to the first dose.
* Febrile illness within 3 days before the first dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
raltegravir AUC and atorvastatin AUC | day 7 of each treatment period
  The comparison of steady state raltegravir (400 mg BID for 7 days) pharmacokinetics (AUC0-12h, Cmax, C12h) with atorvastatin (20 mg QD for 7 days) vs. raltegravir alone by intrasubject comparison.
  The comparison of steady state atorvastatin (20 mg QD for 7 days) pharmacokinetics (AUC0-24h, Cmax, C24h) with raltegravir (400 mg BID for 7 days) vs. atorvastatin alone by intrasubject comparison.

SECONDARY OUTCOMES:
adverse events | entire study
  Adverse events will be scored during the entire study. Laboratory measurements for safety will be collected frequently during the study.
serum LDL cholesterol | Day 1 and day 7 of each treatment period
  12-hour-fasting serum lipid profile (total cholesterol, triglycerides, HDL cholesterol, non-HDL cholesterol, LDL cholesterol) at screening and on the first day and the last day of each treatment period (Days 1, 7, 22, 28, 43 and 49).

CONTACTS AND LOCATIONS:
Overall Officials: David Burger, Principal Investigator — Radboud University Medical Center
Locations (1):
- CRCN Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Result] Blonk M, van Beek M, Colbers A, Schouwenberg B, Burger D. Pharmacokinetic Drug-Drug Interaction Study Between Raltegravir and Atorvastatin 20 mg in Healthy Volunteers. J Acquir Immune Defic Syndr. 2015 May 1;69(1):44-51. doi: 10.1097/QAI.0000000000000544. PMID 25942458
- See also: published results AVIATOR trial — http://www.ncbi.nlm.nih.gov/pubmed/25942458